CLINICAL TRIAL: NCT06117202
Title: The Effect of Interactive Music Therapy Applied for Women During the Perioperative Period for In Vitro Fertilization(IVF) on Their Stress Levels
Brief Title: The Effect of Interactive Music Therapy Applied for Women During the Perioperative Period for IVF on Their Stress Levels
Acronym: IVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Gizem Nur BAYRAM, research assistant doctor, Uludag University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Uludag University1
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy (Experimental): The patients involved in the study will be randomly divided into two groups. One group will be provided with a set of headphones that completely cover the ears and will be played their selected music from a predetermined album for 20 minutes before the procedure. The music will continue to be played through the headphones during the procedure.
  Interventions: Other: music therapy
- control group (No Intervention): The control group will be taken to the operating room with standard anesthesia care protocol.

INTERVENTIONS:
Other: music therapy — The research is a thesis study aimed at determining the stress and anxiety levels of patients seeking in vitro fertilization, investigating influencing factors, and revealing the impact of pre-procedural music listening on these stress and anxiety levels.
  Arms: music therapy

SUMMARY:
The purpose of this study is to investigate the effect of music therapy on stress levels in female patients applying for in vitro fertilization.

DETAILED DESCRIPTION:
If the patients participate in the study, when they apply to the in vitro fertilization center, they will meet with their anesthesiologist, anesthesia assessment will be done face to face and asked some questions about the diseases that may affect the procedure. . If patients are included in the study, their blood pressure, blood oxygen value and heart rate will be measured and recorded, as in every patient. Subsequently, a test will be administered to assess stress and anxiety levels of the patients. The patients involved in the study will be randomly divided into two groups. One group will be provided with a set of headphones that completely cover the ears and will be played their selected music from a predetermined album for 20 minutes before the procedure. The music will continue to be played through the headphones during the procedure. The other group will be taken to the operating room without any procedure, and this process will be applied to both groups. When patients are brought to the operating room, blood pressure, blood oxygen levels, and heart rate will be measured and recorded once again. Routine anesthesia procedures, applicable to all, will be carried out. After patients are fully awake, their pain condition will be assessed using a visual test.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* American Society of Anesthesiologists (ASA) scores I-III.

Exclusion Criteria:

* Patients who did not provide informed consent,
* Used anxiolytics, alcohol, or drugs before the procedure,
* Refused to participate in the study,
* Lost their hearing ability for any reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be conducted on female patients applying to Uludağ University In Vitro Fertilization Unit.
Enrollment: 240 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-03-18 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
stress,anxiety levels | 30 minutes
  The stress levels of the participants will be assessed using the State-Trait Anxiety Inventory scale. The obtained scores theoretically range between 20 and 80. A high score represents a high level of anxiety, while a low score indicates a low level of anxiety.

SECONDARY OUTCOMES:
Postoperative pain level | 30 minutes
  The participants' pain levels will be assessed using the Visual Analog Scale (0-10 point). A score of zero on this scale represents a pain-free condition for the patient, while the highest score reflects the most severe pain they have experienced in their life.

CONTACTS AND LOCATIONS:
Overall Officials: Selcan AKESEN, Study Director — Uludag University
Locations (1):
- Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No